CLINICAL TRIAL: NCT00001400
Title: Outpatient Evaluation of Patients With Known or Suspected Heart Disease (Screening Protocol)
Brief Title: Outpatient Evaluation of Patients With Known or Suspected Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940045; 94-H-0045
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2001-12

CONDITIONS: Heart Disease
Keywords: Heart Disease; Screening; Follow-Up
MeSH Terms: conditions — Heart Diseases

SUMMARY:
This study is designed to screen patients with heart diseases who may qualify to participate in other research studies being conducted by the Cardiology Branch of the National Heart, Lung, and Blood Institute (NHLBI).

Patients participating in this research study will be seen on an outpatient basis and undergo a general medical evaluation, including blood tests, urine, examination, chest x-ray and electrocardiogram (EKG). In addition, patients may be asked to have an echocardiogram (ultrasound scan of the heart) and to perform an exercise stress test.

Patients participating in this study will not receive any investigational treatments.

DETAILED DESCRIPTION:
This protocol permits outpatient screening of patients with cardiovascular diseases who may be candidates for participation in current Cardiology Branch research protocols. No investigational treatments will be administered on this protocol.

ELIGIBILITY:
Must not be enrolled in an active Cardiology Branch research protocol.

The patient must be of scientific interest to the Cardiology Branch, as determined by the investigator.

Patient is being screened for participation in an active protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-12; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States